CLINICAL TRIAL: NCT05832320
Title: Optimum Induction Therapy of Low-risk Acute Promyelocytic Leukemia With All Oral Drugs
Brief Title: Optimum Induction Therapy of Low-risk APL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Xiaolu, Physician-in-charge, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDL 2022-05
Record Dates: First submitted 2023-04-02; First posted 2023-04-27 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Acute Promyelocytic Leukemia; Induction Therapy; Oral
Keywords: Acute Promyelocytic Leukemia; low risk; induction therapy; etoposide
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Etoposide; Tretinoin; Daunorubicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral etoposide with dual induction of ATRA and RIF (Experimental): RIF: 60mg/kg qd, ATRA: 25mg/m2 qd, till CR. When WBC>4.0×109/L, patients will be given oral etoposide (50mg qd to 50mg tid). Cumulative dosage of etoposide during induction ≤1500mg.
  Interventions: Drug: Etoposide
- Daunorubicin with dual induction of ATRA and RIF (Active Comparator): RIF: 60mg/kg qd, ATRA: 25mg/m2 qd, till CR. When WBC>4.0×109/L, patients will be given daunorubicin (20 to 40mg per dose).
  Interventions: Drug: Daunorubicin

INTERVENTIONS:
Drug: Etoposide — Introduction: RIF: 60mg/kg qd, ATRA: 25mg/m2 qd, till CR. When WBC>4.0×109/L, patients will be given oral etoposide (50mg qd to 50mg tid). Cumulative dosage of etoposide during induction ≤1500mg.
  Other Names: all-trans retinoic acid; realgar-indigo naturalis formula
  Arms: Oral etoposide with dual induction of ATRA and RIF
Drug: Daunorubicin — Introduction: RIF: 60mg/kg qd, ATRA: 25mg/m2 qd, till CR. When WBC>4.0×109/L, patients will be given daunorubicin (20 to 40mg per dose).
  Other Names: all-trans retinoic acid; realgar-indigo naturalis formula
  Arms: Daunorubicin with dual induction of ATRA and RIF

SUMMARY:
Despite the high cure probability for acute promyelocytic leukemia (APL), a minority of patients will relapse and the risk factors for relapse are unclear. The goal of this clinical trial is to compare the effectiveness and safety of induction of oral all-trans retinoic acid (ATRA) and realgar-indigo naturalis formula (RIF) combined with oral etoposide or daunorubicin as cytoreductive therapies in low-risk APL. The present study was to explored a cytoreduction of an oral etoposide for low-risk APL with dual induction of ATRA and RIF as a high efficacy, low recurrence, and more convenient all-oral regimen.

DETAILED DESCRIPTION:
Despite the high cure probability for low-risk acute promyelocytic leukemia (APL) in the all-trans retinoic acid (ATRA) era, several clinical problems lead to treatment failure, including early death (ED) and relapse. Previously studies by our group and others showed a relapse of 1.0-4.8% for low-risk APL, and the median time to hematological relapse was 20.5 months after a hematological complete remission (CR). Dur to the largely unclear mechanisms of relapse, the investigators previously explored that a drop of promyelocytic leukemia retinoic acid receptor alpha (PML-RARA) transcript level at the end of induction therapy was associated with a subsequent risk of relapse. The investigators and others have indicated that the addition of cytarabine in induction therapy might correlate with lower relapse rate. Whether cytoreduction in induction therapy has prognostic significance in APL, besides its role in leukocytosis, remains unclear. Etoposide is a topoisomerase II inhibitor antitumor agent which is widely used in the treatment of several hematological malignancies. The successful experience in high-risk APL demonstrated the efficacy, safety and convenience of oral etoposide as an alternative cytoreductive agent at the initial stage of induction therapy. Therefore, the present prospective study is conducted to explore the potential role of cytoreduction during induction therapy on prognosis, and further exploit the all-oral induction regimen for low-risk APL with etoposide combined with ATRA plus RIF as the front-line therapy for low-risk APL.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed APL patients (WHO 2008 diagnostic classification);
* 18-75 years old;
* Liver function: propionate hydrogentransferase (ALT) and aspartate hydrogentransferase (AST) ≤ 2.5 times the upper limit of normal value, bilirubin ≤ 2 times the upper limit of normal value;
* Renal function: muscle salt ≤ 3 times the upper limit of normal value;
* The physical strength score is 0-2 (ECOG);
* White blood cells ≤ 10×109/L;
* Subjects must sign an informed consent form.

Exclusion Criteria:

* Subjects who have participated in other clinical trials within 30 days;
* Pregnant and lactating subjects;
* Subjects who are known to be HIV-positive in serological tests;
* Subjects who have viral hepatitis serological test positive;
* Subjects who have severe arrhythmia, abnormal electrocardiogram (QT>500ms);
* Subjects who suffer from mental illness or unable to cooperate with the research treatment and monitoring requirements due to other diseases;
* Subjects who participate in other clinical research at the same time;
* Subjects who fail to sign the informed consent form;
* Other conditions that the researchers think are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission | At the end of induction therapy within 45 days after diagnosis
  Haematological CR was defined as a proportion of BM blasts of <5%, the absence of blasts in Auer rods, the absence of extramedullary disease, an absolute neutrophil count of >1×10⁹/L and a platelet count of >100×109/L, with no red-cell transfusions
Promyelocytic leukaemia-retinoic acid receptor alpha (PML-RARA) transcript levels of ≥6.5% at the end of induction therapy | At the end of induction therapy within 45 days after diagnosis
  PML-RARA transcripts using Abelson tyrosine-protein kinase (ABL) as an internal control by quantitative RT-PCR

SECONDARY OUTCOMES:
Early death (ED) | During the induction therapy within 30 days after diagnosis
  Defined as death within 30 days after diagnosis
Cumulative recurrence rate | From date of randomization until the date of last documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  A measure of the total relapse that a certain event will happen during a given period of time
2-year event-free survival rate | From the time of randomization to the time of last follow-up within 2 years after diagnosis
  The EFS was defined as the time from diagnosis to the following events: no haematological CR after induction therapy; no CMR after consolidation therapy, molecular relapse, haematological relapse; death from any cause; or last follow-up.
Satefy. Common haematological and non-haematological adverse events were monitored twice per week during induction and twice per month during consolidation. | From the time of randomization to the time of last follow-up within 2years after diagnosis
  Toxic effects were graded according to the 'WHO classification standard for acute and subacute toxicity of anticancer drugs'.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolu Zhu, Doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No